CLINICAL TRIAL: NCT06371690
Title: The Effects of Using the Web-Based Double Eye Control Program on Medication of High Risk Drugs in Pediatric Patients: The Effect of Web-Based Double Eye Control Program
Brief Title: The Effects of Using the Web-Based Double Eye Control Program on Medication Error
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Ege University (Other)
Responsible Party: Principal Investigator, Beste Ozguven Oztornaci, Assistant Professor Doctor, Izmir Katip Celebi University
Other Study IDs: 17-11/37
Record Dates: First submitted 2023-12-30; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Main Heading (Descriptor) Terms
Keywords: Child; Child Nursing; High-Risk Drugs; Medication Error; Error Prevention Strategies

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Medication errors during the application of high-risk drugs: Medication Errors During the Application of High-risk Drugs Before and After Using Web-Based Double-Eye Control Program
  Interventions: Other: Web-Based Double-Eye Control Program

INTERVENTIONS:
Other: Web-Based Double-Eye Control Program — Web-Based Double-Eye Control Program, a web-based drug dose calculation program, is compatible with smartphones, tablets and computers. On the interface of the website, the nurse is required to enter data such as the age, weight, medications and doses ordered by the physician of the patient. When all these data are entered, the amount of medication that the nurse should give and whether the ordered dose is within the safe dose range for the patient are calculated by the program, so that the nurse can control her own calculations. On the other interface of the website, there are medication instructions uploaded by the researchers. With this interface, nurses access all pharmacological information about especially high-risk drugs (indications, contraindications, interacting drugs and fluids, fluids to be used for diluting, medication route, medication pace, etc.) and information that will enable the medication to be carried out in a standard way.

SUMMARY:
Methods: The study was carried out as a quasi-experimental study in the Pediatric Surgery Clinics of a university hospital using the "Pre-Test-Post-Test Model in a Single Group". The sample of the study consisted of all high-risk drugs administered by 24 nurses working in these clinics, taking part in medication and agreeing to take part in the study. Data were collected by the researcher using the Medication Observation Form. The Form was created based on the literature, and by making use of the "10 Correct Rules in Medication" and the Medication Skills Steps in the Double Eye Control Program. In the first step, medication error rates were determined through observation method. In the second step; the Web-Based Double-Eye Control Program, which is a standard drug dose calculation and medication program created by the researchers, was started to be implemented. Medication error rates were determined again through post-intervention observation method. Informed voluntary consent, ethics committee and hospital permissions were obtained for the implementation of the study.

DETAILED DESCRIPTION:
Background: In this study, it was aimed to examine the effect of using Web Based Double-Eye Control Program as a new decision support system in preventing errors and standardization in high-risk medications of pediatric nurses.

Methods: The study was carried out as a quasi-experimental study in the Pediatric Surgery Clinics of a university hospital using the "Pre-Test-Post-Test Model in a Single Group". The sample of the study consisted of all high-risk drugs (532 before the intervention, 538 after the intervention, a total of 1070 drug doses) administered by 24 nurses working in these clinics, taking part in medication and agreeing to take part in the study. Data were collected by the researcher using the Medication Observation Form. The Form was created based on the literature, and by making use of the "10 Correct Rules in Medication" and the Medication Skills Steps in the Double Eye Control Program. In the first step, medication error rates were determined through observation method. In the second step; the Web-Based Double-Eye Control Program, which is a standard drug dose calculation and medication program created by the researchers, was started to be implemented. Medication error rates were determined again through post-intervention observation method. Informed voluntary consent, ethics committee and hospital permissions were obtained for the implementation of the study.

ELIGIBILITY:
Inclusion Criteria:

* The medications observed were to be in the high-risk drug group for children,
* Volunteering of nurses working in the clinic to participate in the research,
* Nurses working in the clinic should have had proper level of internet usage knowledge to use a web-based program.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of the research was composed of Nurses working in the Pediatric Surgery Department Clinic (Pediatric Surgery, Pediatric Surgery Intensive Care, Neonatal Surgery Intensive Care Clinics) of a university hospital in Turkey between November 2017 and June 2018, and all high-risk drugs they administered.
Sampling Method: Non-Probability Sample
Enrollment: 1070 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Error rates | Between January 2017 and September 2018
  Medication errors during administration of high-risk drugs in pediatric patients

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University, Izmir, Çi̇ğli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided